CLINICAL TRIAL: NCT03720184
Title: Haemo-autologous Antegrade Repriming (HAR) Clinical Trial for Validation as Minimum Impact Perfusion Strategy in Cardiopulmonary Bypass
Brief Title: Haemo-autologous Antegrade Repriming (HAR) as Minimum Impact Perfusion Strategy for Cardiopulmonary Bypass
Acronym: HARjbm1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Juan Blanco Morillo (Other)
Collaborators: Instituto Murciano de Investigación Biosanitaria Virgen de la Arrixaca (Other)
Responsible Party: Sponsor-Investigator, Juan Blanco Morillo, Principal Investigator, Hospital Universitario Virgen de la Arrixaca
Organization: Hospital Universitario Virgen de la Arrixaca (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HARjbm1
Record Dates: First submitted 2018-10-18; First posted 2018-10-25 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Anemia; Cognitive; Disorder, Due to General Medical Condition; Embolism, Air; Transfusion; Cardiac Disease; Extracorporeal Circulation; Complications; Valve Anomalies
Keywords: Retrograde autologous priming; RAP; HAR; cardiopulmonary bypass; Extracorporeal circulation; Gaseous microemboli; perfusion
MeSH Terms: conditions — Anemia; Embolism, Air; Heart Diseases

STUDY DESIGN:
Intervention Model Description: In a preliminary phase, patients are randomly assigned to 4 branches, regarding to two conditions: oxygenator´s deairing type and HAR exposure. This phase is designed as pilot study with 100 patients in order to determine precisely the sample size needed depending on the observed effects.
  If there are no clinical differences between oxygenators behaviour, during the second stage, sample will be only divided in 2 groups due to HAR exposure.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patient and neurocognitive examinator does not know the arm assigned, as well as the anaesthesiologist, surgeon and ICU team. Only the perfusionist has access to de randomization sheet before choosing and set up of the extracorporeal circuit.
  In order to guarantee the blinding, the perfusionist must be hidden during the possible HAR performance, using a field blanket to isolate the oxygenator´s area. Anestesiologist´s proceed in every case as if HAR is assigned maintaining a mean arterial pressure over 60 mmHg.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAR group (Experimental): Treated group is exposed to an haematic antegrade autologous repriming of the MiECC CLass IV circuit, reducing the haemodilution related to CPB initiation to a fix amount of 300ml
  Interventions: Procedure: HAR
- Control Group (No Intervention): Control group is not exposed to HAR. The extracorporeal circuit is a MiECC primed with 1000ml of Isofundin (crystalloid balanced solution) as an standard circuit

INTERVENTIONS:
Procedure: HAR — HAR, the 6 steps procedure that results in 300ml of haemodilution. Step 0: Circuit is primed with 1000ml of crystalloid solution. Step 1: Venous line content is drained to the reservoir. Step 2: arterial srystalloid priming is displaced to the reservoir retrogradely by autologous blood. Step 3: Crystalloid priming is discarded to the collector bag. Step 4: An amount of 300ml of arterial blood is sequestered to the reservoir avoiding the mixture. Step 5: The centrifugal pump and the oxygenator are reprimed with autologous blood displacing the priming and GME to the collector bag. Step 6: CPB is initiated with a low haemodilution of 300ml.
  Available at: https://zenodo.org/record/4276132#.X7K8AchKgRk
  Other Names: Haematic antegrade repriming; Extracorporeal circuit repriming
  Arms: HAR group

SUMMARY:
Haemo-autologous Antegrade Repriming (HAR) is a procedure based in the combination of evidence proven measures designed to reduce the haemodilution caused by establishing the cardiopulmonary bypass (CPB) during cardiac surgery.

This clinical trial aims to determinate, in one hand, the benefits related to HAR in terms of transfusion, ICU stay, ventilation time, early mortality and complications. In the other hand analyzes the gaseous microemboli (GME) load, comparing the oxygenators venting technology´s efficiency in treatment and control group, and its relation with patient´s neurocognitive status.

DETAILED DESCRIPTION:
HAR is a repriming technique based in Retrograde Autologous Priming (RAP), that has been implemented by recently recommended measures in terms of reducing blood transfusions.

The expected clinical benefits are related to hemodilution´s reduction up to only 300ml. The extracorporeal circuit has been reduced to 3/8 inch diameter in both lines, reducing the surface up to 1000ml of dynamic priming.

Vacuum assisted venous drainage (VAVD) allows to empty the venous line after priming and deairing, facilitating the venous flow for CPB initiation.

The antegrade repriming eliminates the maximum amount of crystalloid contained in the circuit, displacing it to a collector bag, by using autologous blood sequestered from the arterial line to the hardshell reservoir.

HAR reduces the CPB hemodilution related to priming from 1500 to 300 ml preventing the usual sudden haemoglobin level reduction occured during every extracorporeal techinque´s establishment.

Our mission is to analyze if HAR can be validated as a safe and effective tool to improve clinical outcomes in cardiac surgery procedures under extracorporeal circulation

ELIGIBILITY:
Inclusion Criteria:

- All patients purposed to undergo elective cardiopulmonary bypass for cardiac valve surgery or other pathologies requiring to open heart chambers.

Exclusion Criteria:

* Urgency and emergency
* Heart transplantations
* Severe cognitive affection
* Active sepsis
* Previous anemia
* Early re-intervention
* Pre-Op extracorporeal membrane oxygenation (ECMO) support
* Hemodynamic unstability during HAR
* Any clinical condition that may force protocol deviation

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2021-02-09 (Actual)

PRIMARY OUTCOMES:
Transfusion | 1 year
  Blood product consumption during patients hospital stay
ICU stay | 1 year
  Length of stay at Intensive Care Unit. (days)
Ventilation time | 1 year
  Hours under mechanical ventilation after surgery
Complications | 1 year
  Incidence of neurological, respiratory, urinary, cardiologic complications and multiorganic failure
Mortality | 1 year
  Incidence of death during hospital stay

SECONDARY OUTCOMES:
Emboli number | 1 year
  Number of total gaseous microemboli delivered by the extracorporeal system to the patient
Emboli Volume | 1 year
  Volume of total gaseous microemboli delivered by the extracorporeal system to the patient
Emotional regulation | 6 months after surgery
  Evolution of Emotional regulation test results, comparing the variation with the amount of embolic events detected during the extracorporeal procedure. (4-6 months)
Visual work memory variation and emboli | 6 months after surgery
  Evolution of Visuospatial working memory test results, comparing the variation of the basal status and short term measurements (4-6 months after surgery) with the amount of detected emboli delivered to the patient through the heart-lung machine´s circuit.
Executive functions and emboli | 6 months after surgery
  Analysis of the clock drawing test variation, comparing basal and short term (4-6 months after surgery) measurements, and the expected relation with the emboli detected during the extracorporeal technique
Visual memory and cognitive status evaluation and emboli | 6 months after surgery
  Analysis of the variation of cognitive functions using picture tests(comparing basal status and short term evaluation results (4-6 months after surgery) and the amount of emboli delivered to the patient during the cardiopulmonary bypass

CONTACTS AND LOCATIONS:
Overall Officials: Juan B Morillo, M.Sc, Principal Investigator — IMIB. University Hospital Virgen de la Arrixaca. Murcia
Locations (1):
- Hospital Clinico universitario Virgen de la Arrixaca, Murcia, MU, Spain

REFERENCES:
- [Background] Loor G, Rajeswaran J, Li L, Sabik JF 3rd, Blackstone EH, McCrae KR, Koch CG. The least of 3 evils: exposure to red blood cell transfusion, anemia, or both? J Thorac Cardiovasc Surg. 2013 Dec;146(6):1480-1487.e6. doi: 10.1016/j.jtcvs.2013.06.033. Epub 2013 Aug 30. PMID 23998782
- [Background] Liu YH, Wang DX, Li LH, Wu XM, Shan GJ, Su Y, Li J, Yu QJ, Shi CX, Huang YN, Sun W. The effects of cardiopulmonary bypass on the number of cerebral microemboli and the incidence of cognitive dysfunction after coronary artery bypass graft surgery. Anesth Analg. 2009 Oct;109(4):1013-22. doi: 10.1213/ane.0b013e3181aed2bb. PMID 19762724
- [Background] Wang S, Undar A. Vacuum-assisted venous drainage and gaseous microemboli in cardiopulmonary bypass. J Extra Corpor Technol. 2008 Dec;40(4):249-56. PMID 19192754
- [Background] Evered L, Scott DA, Silbert B, Maruff P. Postoperative cognitive dysfunction is independent of type of surgery and anesthetic. Anesth Analg. 2011 May;112(5):1179-85. doi: 10.1213/ANE.0b013e318215217e. Epub 2011 Apr 7. PMID 21474666
- [Background] Zhang X, Yan X, Gorman J, Hoffman SN, Zhang L, Boscarino JA. Perioperative hyperglycemia is associated with postoperative neurocognitive disorders after cardiac surgery. Neuropsychiatr Dis Treat. 2014 Feb 19;10:361-70. doi: 10.2147/NDT.S57761. eCollection 2014. PMID 24570589
- [Background] Segers T, Stehouwer MC, de Somer FMJJ, de Mol BA, Versluis M. Optical verification and in-vitro characterization of two commercially available acoustic bubble counters for cardiopulmonary bypass systems. Perfusion. 2018 Jan;33(1):16-24. doi: 10.1177/0267659117722595. Epub 2017 Aug 2. PMID 28766987
- [Background] Lazar RM, Pavol MA, Bormann T, Dwyer MG, Kraemer C, White R, Zivadinov R, Wertheimer JC, Thone-Otto A, Ravdin LD, Naugle R, Mechanic-Hamilton D, Garmoe WS, Stringer AY, Bender HA, Kapadia SR, Kodali S, Ghanem A, Linke A, Mehran R, Virmani R, Nazif T, Parhizgar A, Leon MB. Neurocognition and Cerebral Lesion Burden in High-Risk Patients Before Undergoing Transcatheter Aortic Valve Replacement: Insights From the SENTINEL Trial. JACC Cardiovasc Interv. 2018 Feb 26;11(4):384-392. doi: 10.1016/j.jcin.2017.10.041. Epub 2018 Feb 1. PMID 29397361
- [Background] Kurusz M, Butler BD. Bubbles and bypass: an update. Perfusion. 2004;19 Suppl 1:S49-55. doi: 10.1191/0267659104pf720oa. PMID 15161064
- [Result] Vandewiele K, Bove T, De Somer FM, Dujardin D, Vanackere M, De Smet D, Moerman AT, Bouchez S, Francois K. The effect of retrograde autologous priming volume on haemodilution and transfusion requirements during cardiac surgery. Interact Cardiovasc Thorac Surg. 2013 Jun;16(6):778-83. doi: 10.1093/icvts/ivt085. Epub 2013 Mar 12. PMID 23482374
- [Result] Spellman T, Rigotti M, Ahmari SE, Fusi S, Gogos JA, Gordon JA. Hippocampal-prefrontal input supports spatial encoding in working memory. Nature. 2015 Jun 18;522(7556):309-14. doi: 10.1038/nature14445. Epub 2015 Jun 8. PMID 26053122
- [Result] De Somer FM, Vetrano MR, Van Beeck JP, Van Nooten GJ. Extracorporeal bubbles: a word of caution. Interact Cardiovasc Thorac Surg. 2010 Jun;10(6):995-1001. doi: 10.1510/icvts.2009.229088. Epub 2010 Mar 2. PMID 20197351
- [Result] Basciani R, Kroninger F, Gygax E, Jenni H, Reineke D, Stucki M, Hagenbuch N, Carrel T, Eberle B, Erdoes G. Cerebral Microembolization During Aortic Valve Replacement Using Minimally Invasive or Conventional Extracorporeal Circulation: A Randomized Trial. Artif Organs. 2016 Dec;40(12):E280-E291. doi: 10.1111/aor.12744. Epub 2016 Jun 10. PMID 27283935
- [Result] Abrahamov D, Levran O, Naparstek S, Refaeli Y, Kaptson S, Abu Salah M, Ishai Y, Sahar G. Blood-Brain Barrier Disruption After Cardiopulmonary Bypass: Diagnosis and Correlation to Cognition. Ann Thorac Surg. 2017 Jul;104(1):161-169. doi: 10.1016/j.athoracsur.2016.10.043. Epub 2017 Feb 10. PMID 28193536
- [Result] Society of Thoracic Surgeons Blood Conservation Guideline Task Force; Ferraris VA, Brown JR, Despotis GJ, Hammon JW, Reece TB, Saha SP, Song HK, Clough ER; Society of Cardiovascular Anesthesiologists Special Task Force on Blood Transfusion; Shore-Lesserson LJ, Goodnough LT, Mazer CD, Shander A, Stafford-Smith M, Waters J; International Consortium for Evidence Based Perfusion; Baker RA, Dickinson TA, FitzGerald DJ, Likosky DS, Shann KG. 2011 update to the Society of Thoracic Surgeons and the Society of Cardiovascular Anesthesiologists blood conservation clinical practice guidelines. Ann Thorac Surg. 2011 Mar;91(3):944-82. doi: 10.1016/j.athoracsur.2010.11.078. PMID 21353044
- See also: To assess and compare the effectiveness and costs of Phototest,Screen for dementia (DEM) and cognitive impairment (CI). — https://doi.org/10.1186/1471-2377-11-92
- See also: Effect of blood transfusion on long-term survival after cardiac operation — http://linkinghub.elsevier.com/retrieve/pii/S0003497502037669